CLINICAL TRIAL: NCT07356921
Title: Function of Ligamentum Teres in Management of Developmental Hip Dysplasia (DDH)
Brief Title: Ligamentum Teres in Management of Developmental Hip Dysplasia
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Bahaaeldin Mohamed Abdelhafez, Principal Investigator, Assiut University
Other Study IDs: LTDDH
Record Dates: First submitted 2026-01-13; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Orthopaedic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: ligamentum teres tenodesis — * Creating a tract or tunnel: from acetabulum cavity to intra pelvic cavity using bit (3.5mm or 4.5mm according to the size of the ligament) or k wire (3mm) from the site of the ligamentum attached at the acetabulum guided with passer
  * Passing of the sutured ligamentum teres through the tunnel
  * Tighting of the passed sutured ligamentum teres

SUMMARY:
Treatment of developmental dysplasia of the hip (DDH) is still challenging, till now there is no any recent advances have refined our understanding of how best to survey for the condition during infancy and refine the selection of patients who can best benefit from hip preservation surgery.

DETAILED DESCRIPTION:
Concentric positioning of femoral head into the acetabular cavity and adequate balance in growth between tri-radiate and acetabular cartilage are leading to adequate growth and development of the hip. Any alteration in these two conditions leads to a hip dysplasia & dislocation .

Treatment of developmental dysplasia of the hip (DDH) is still challenging, till now there is no any recent advances have refined our understanding of how best to survey for the condition during infancy and refine the selection of patients who can best benefit from hip preservation surgery.

The ideal continued target would be to prevent missed hip dislocations or dysplasia during the infant period, decrease the incidence of total hip arthroplasty in adulthood related to undertreat DDH and prevent avascular necrosis (AVN).

The goal of the treatment is to achieve a concentric reduction of the femoral head into the acetabulum.

ELIGIBILITY:
Inclusion Criteria:

* Virgin developmental dysplasia of the hip (DDH)
* failed closed reduction in the management of DDH and failed open reduction through medial approach in the management of DDH

Exclusion Criteria:

* cases that managed previously through anterior approach
* old neglected cases above 5 years old children

Ages: 9 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Operation was done under general anesthesia and patient in supine position. Sterilization was done. Incision was made from anterior half of iliac crest to ASIS (the anterior or anterolateral Smith-Petersen approach with a modified "bikini" incision) .Superficial dissection was done by identify gap between sartorius and tensor fasciae latae, dissect through subcutaneous fat (avoid lateral femoral cutaneous n.), incise fascia on medial side of tensor fascia latae and detach origin of tensor fasciae latae of iliac to develop internervous plane. Deep dissection was done by identify plane between rectus femoris and gluteus medius and detaches rectus femoris from both its origins.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
modified Harris Hip Score | 6 months

REFERENCES:
- [Background] Bache CE, Graham HK, Dickens DR, Donnan L, Johnson MB, Nattrass G, O'Sullivan M, Torode IP. Ligamentum teres tenodesis in medial approach open reduction for developmental dislocation of the hip. J Pediatr Orthop. 2008 Sep;28(6):607-13. doi: 10.1097/BPO.0b013e318184202c. PMID 18724195
- [Background] Wenger DR, Mubarak SJ, Henderson PC, Miyanji F. Ligamentum teres maintenance and transfer as a stabilizer in open reduction for pediatric hip dislocation: surgical technique and early clinical results. J Child Orthop. 2008 Jun;2(3):177-85. doi: 10.1007/s11832-008-0103-3. Epub 2008 Apr 29. PMID 19308575